CLINICAL TRIAL: NCT00995319
Title: Acute and Longlasting Side Effects Caused by Radiotherapy in the Head and Neck Area
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Other Study IDs: 17436
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Head and Neck Cancer
Keywords: mouth; Mucositis; Dysphagia; malnutrition; Xerostomia; saliva; tooth injuries
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Deglutition Disorders; Malnutrition; Xerostomia; Tooth Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- radiation patients: cancer patients with radiotherapy concerning the head and neck area/oral cavity

SUMMARY:
The purpose of this clinical investigation is to evaluate acute and longlasting side effects in patients undergoing radiotherapy for cancer treatment in the head and neck area.

DETAILED DESCRIPTION:
The "Dental Team" at the Department for Oral and Maxillofacial Surgery in Trondheim takes care of patients before, during and also after radiotherapy in the head and neck area. In spite of the use of advanced radiation protocols and prevention measures such as fluoridation splints the team observes significant side effects, both under radiation and also on the long term after concluding treatment. Common problems are for example dermal and mucosal damages, reduced salivation, dysphagia and lesions of the teeth. Aim of the study is the investigation and documentation of side effects and complications in relation to the oral cavity. During the acute and postradiation phase a continuous follow-up over a longer lasting period is proceeded with registration of all relevant parameters. This includes among others dental status and evaluation of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* radiation concerning the oral cavity
* follow-up at the Dental Team

Exclusion Criteria:

* refused approval
* survival prognosis under one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cancer patients with radiation therapy concerning the oral cavity who are in care of the Detal Team at St.Olavs University Hospital
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
salivary flow | 3 months
salivary flow | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph M Ziegler, Prof.Dr.Dr., Study Director — St.Olavs Hospital / NTNU
Locations (1):
- Department for Oral and Maxillofacial Surgery, St.Olavs Hospital / NTNU, Trondheim, Norway